CLINICAL TRIAL: NCT01872663
Title: Influence of Different Physical Therapy Resources Application After Abdominal Surgery
Brief Title: Influence of Different Physical Therapy Resources Application After Reduction Stomach Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Eli Maria Pazzianotto Forti, PhD, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Patricia2013; UNIMEP2013 (Other: UNIMEP)
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Pulmonary Atelectasis; Respiratory Tract Diseases; Pathological Conditions, Signs and Symptoms
Keywords: Morbid obesity; Bariatric surgery; Pulmonary atelectasis; Spirometry; Continuos Positive Airway Pressure; Physical therapy speciality
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Tract Diseases; Pathological Conditions, Signs and Symptoms; Obesity, Morbid | interventions — Continuous Positive Airway Pressure; Intermittent Positive-Pressure Breathing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Incentive spirometry (Voldyne®) (Experimental): Individuals will be treated with incentive spirometry, Voldyne Model 5000® in the immediate and the first postoperative day, twice a day, in sessions of 6 sets of 15 repetitions each, with an interval of four hours between them.
  Interventions: Procedure: Incentive spirometry
- Continuous positive airway pressure (Experimental): Individuals will be treated with flow generator(Whisperflow, Caradyne, Ireland)and valve PEEP type spring-loaded which remain 10 cmH2O, in the immediate and the first postoperative day, twice a day, in sessions 30 minutes each, with an interval of four hours between them.
  Interventions: Procedure: Continuous positive airway pressure; Procedure: Expiratory Positive Airway Pressure
- Expiratory Positive Airway Pressure (Experimental): Subjects will be treated with oronasal mask affixed to the face, with the PEEP valve set at 10 cmH2O, in the immediate and the first postoperative day, twice a day, in sessions of 6 sets of 15 repetitions each, with an interval of four hours between them.
  Interventions: Procedure: Continuous positive airway pressure; Procedure: Expiratory Positive Airway Pressure
- Intermittent positive pressure breathing (Experimental): Subjects will be treated with application of Müller Resuscitator (Engesp®) through a nozzle, using a pressure endotracheal 20-30 cmH2O, refering to 2-3 kgf/cm², adjusted throttle valve oxygen, according to the patient's comfort and the micronebulizer coupled only saline as the diluent. The procedure will be performed in the immediate and the first postoperative day, twice a day, in sessions of 6 sets of 15 repetitions each, with an interval of four hours between them.
  Interventions: Procedure: Continuous positive airway pressure; Procedure: Intermittent positive pressure breathing
- Bi-level positive airway pressure (Experimental): Individuals will be treated with positive pressure in the BiPAP mode (Bi-level positive airway pressure) in the immediate and the first postoperative day, twice a day, in sessions 30 minutes each, with an interval of four hours between them.
  Interventions: Procedure: Continuous positive airway pressure; Procedure: Expiratory Positive Airway Pressure; Procedure: Bi-level positive airway pressure
- Breath Stacking (Experimental): Subjects will be treated with a siliconized mask connected to a unidirectional valve and adapted to the patient's face, allowing only the inspiration and the expiratory limb remains occluded, while the volunteer is instructed to perform successives inspiratory efforts, in the immediate and the first postoperative day, twice a day, in sessions of 6 sets of 15 repetitions each, with an interval of four hours between them.
  Interventions: Procedure: Breath Stacking
- Control (No Intervention): Individuals will be treated with conventional physiotherapy according to the routine service of physiotherapy of the hospital.

INTERVENTIONS:
Procedure: Continuous positive airway pressure — The use of positive pressure airway seeking the prevention or treatment of hypoxic respiratory failure, improved arterial oxygenation, restoration or maintenance of lung volume reduction and atelectasis, decrease the work of breathing, decreased dyspnea index and increased residual volume.
  Arms: Bi-level positive airway pressure; Continuous positive airway pressure; Expiratory Positive Airway Pressure; Intermittent positive pressure breathing
Procedure: Incentive spirometry — The volume of incentive spirometry (Voldyne ®) is able to provide increased transpulmonary pressure gradient, which can prevent or reverse atelectasis.
  Arms: Incentive spirometry (Voldyne®)
Procedure: Breath Stacking — The method allowed to obtain a maximum lung expansion with minimal patient compliance.
  Arms: Breath Stacking
Procedure: Expiratory Positive Airway Pressure — The use of positive pressure airway seeking the prevention or treatment of hypoxic respiratory failure, improved arterial oxygenation, restoration or maintenance of lung volume reduction and atelectasis, decrease the work of breathing, decreased dyspnea index and increased residual volume.
  Arms: Bi-level positive airway pressure; Continuous positive airway pressure; Expiratory Positive Airway Pressure
Procedure: Intermittent positive pressure breathing — The use of positive pressure airway seeking the prevention or treatment of hypoxic respiratory failure, improved arterial oxygenation, restoration or maintenance of lung volume reduction and atelectasis, decrease the work of breathing, decreased dyspnea index and increased residual volume.
  Arms: Intermittent positive pressure breathing
Procedure: Bi-level positive airway pressure — The use of positive pressure airway seeking the prevention or treatment of hypoxic respiratory failure, improved arterial oxygenation, restoration or maintenance of lung volume reduction and atelectasis, decrease the work of breathing, decreased dyspnea index and increased residual volume.
  Arms: Bi-level positive airway pressure

SUMMARY:
The aim of this study will be to investigate the effects of using physical therapy resources in the postoperative morbidly obese individuals undergoing gastroplasty.

It is believed that the application of these various features of physiotherapy after abdominal surgery may contribute differently in restoring lung function and prevention of pulmonary complications and can thus identify the resources that can contribute more effectively in post-operative bariatric surgery.

DETAILED DESCRIPTION:
The aim of this study will be to investigate the effects of using physical therapy resources in the postoperative morbidly obese individuals undergoing Roux-en-Y gastric by-pass with regard to: lung volumes and capacities, prevalence of atelectasis, thoracoabdominal mobility and evaluation of peak flow of cough, evaluated pre and post operative.

Individuals with BMI between 40 and 55 Kg/m², aged between 25 and 55 years, underwent the surgical procedure Roux-en-Y type gastric by-pass by laparotomy and normal preoperative pulmonary function will be included.

The volunteers will be divided into seven different groups, according to the treatment received during hospitalization after surgery:

G control: subjects treated with conventional physiotherapy according to the routine service of physiotherapy of the hospital; G Voldyne: subjects treated with incentive spirometry, Voldyne Model 5000® (Sherwood Medical, USA); G CPAP: subjects treated with "continuous positive airway pressure"; G EPAP: subjects treated with "expiratory positive airway pressure"; G IPPB: subjects treated with "intermittent positive pressure breathing"; G BIPAP: subjects treated with "bi-level positive airway pressure"; G BS: subjects treated with "breath stacking" (siliconized mask connected to a unidirectional valve allowing only inspiration).

The application of resources will be held twice a day in the immediate and in the first postoperative sessions in 6 sets of 15 reps or 30 continuous minutes, with an interval of 4 hours between sessions. The researcher will remain alongside the volunteers, following them and monitoring vital signs and respiratory comfort.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 40 and 55 Kg/m²
* Aged between 25 and 55 years
* Submitted to Roux-en-Y type gastric by-pass by laparotomy
* Normal preoperative pulmonary function test

Exclusion Criteria:

* Hemodynamic instability
* Hospital stay longer than three days
* Presence of postoperative complications
* Smoking

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 2 days after surgery
  Spirometry was carried out according to the guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS) (2005). Three types of maneuver were used in order to evaluate the lung volumes and flows: Slow Vital Capacity (SVC), Forced Vital Capacity (FVC) and Maximum Voluntary Ventilation (MVV). The maneuvers were carried out until three acceptable and reproducible curves were obtained, not exceeding more than eight attempts. The values extracted from each maneuver were selected according to Pereira (2002), and the predicted values calculated using the equation proposed by Pereira et al. (1992) for Brazilians.

SECONDARY OUTCOMES:
Prevalence of atelectasis | 2 days after surgery
  The radiological report on the inspiration radiography, issued by the hospital radiologist, was used to analyze the presence of atelectasis.
Thoracoabdominal mobility | 2 days after surgery
  The measurement of thoracoabdominal mobility was performed by using a tape scaled in centimeters. In the standing position, the measurements were made at levels axillary, xiphoid and abdominal during rest, and at maximal inspiration and maximal expiration. At each level, the measurements were performed three times. It computed the highest value of inspiration and the lowest of expiration. The absolute difference between these values was considered the thoracoabdominal mobility.
Peak cough flow | 2 days after surgery
  The peak flow measured during a cough maneuver will be measured by the equipment Peak Flow ®. For this, the volunteer will be instructed to place the mouthpiece between the lips of the equipment and play a cough with nostrils occluded nose clip. The maneuver should be repeated three times and the best preoperative measures will be compared to the best postoperative measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Metodista de Piracicaba (UNIMEP), Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Brigatto P, Carbinatto JC, Costa CM, Montebelo MI, Rasera-Junior I, Pazzianotto-Forti EM. Application of positive airway pressure in restoring pulmonary function and thoracic mobility in the postoperative period of bariatric surgery: a randomized clinical trial. Braz J Phys Ther. 2014 Nov-Dec;18(6):553-62. doi: 10.1590/bjpt-rbf.2014.0054. Epub 2015 Jan 9. PMID 25590448